CLINICAL TRIAL: NCT02059928
Title: Intraosseous Pressure Monitoring in Intensive Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-149
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-04

CONDITIONS: Blood Pressure
Keywords: fluid resuscitation; invasive pressure monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraosseous device placement (Experimental): Intraosseous device
  Interventions: Device: Intraosseous Device

INTERVENTIONS:
Device: Intraosseous Device
  Other Names: EZ-IO Needle Set and Driver

SUMMARY:
In emergency situations, access to the venous system is essential in order to administer fluids and medication and to monitor patients. When peripheral veins are difficult to access or the patient's condition requires certain medications, or monitoring, central venous catheters (CVC) are inserted. CVC placement introduces a much higher level of risk compared to peripheral catheters. The technique of intraosseous (IO) infusion has been used by healthcare professionals for several decades, but recently has gained wide popularity in the emergency care settings. This technique allows providers to secure a needle in the bony matrix at the ends of long bones (tibia and humerus) and infuse fluids and medications into the intramedullary space. The ability to monitor a patient's blood pressure through an intraosseous needle is unknown. The primary objective of this study is to describe the relationship (ratio) of intraosseous pressure (IOP) values to standard pressure values, including systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), and central venous pressure (CVP).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Admitted to the surgical intensive care units
* Current central pressure monitoring through a central line
* Patient currently intubated and sedated
* Informed consent obtained from family member
* English speaking patient

Exclusion Criteria:

* Known implanted devices in the humerus or tibia that prohibit placement of the intraosseous needle.
* Known osteoporosis, avascular necrosis, or other bone pathology affecting bone healing.
* Fracture or other significant injury to the tibia or humerus or surrounding musculature/tissue.
* Inability to landmark IO placement due to excessive tissue over placement location.
* Anticipated surgery within 12 hours of time of consent
* Current infection at the placement site.
* Previous, significant orthopedic procedure at the site
* Pregnant or has the potential for being pregnant
* Prisoner of the state
* Minor (< 18 years old)
* Inability to obtain informed consent from family member
* Non-English speaking patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J Frascone, MD, Principal Investigator — Regions Hospital; Josh Salzman, MA, Study Director — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intraosseous Device Placement: Intraosseous device
  Intraosseous Device pressure measurement
Period: Overall Study
Arm/Group | Intraosseous Device Placement
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Twenty patients were enrolled between January 2014 and May 2015
Groups:
- Intraosseous Device Placement: Intraosseous device
  Intraosseous Pressure Monitoring in Surgical Intensive Care Unit Patients
Arm/Group | Intraosseous Device Placement
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 60 [45 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Standardized Ratio as a Percentage Between Mean IOP and Mean Arterial Pressure
Description: External cuff pressure readings were recorded every 15 minutes, and IO pressure data obtained via pressure transducer was recorded continuously for up to 12 hours. IO systolic, diastolic, and mean pressure (IO SBP, IO DBP, IO Mean) readings were summarized for the minute before and minute following an external cuff pressure reading. The ratios as a percentage of IO pressures to external cuff pressures (IO Systolic Blood Pressure / Cuff SBP; IO DBP / Cuff DBP; IO Mean / Cuff Mean) were calculated.
Time Frame: Up to 12 hour data collection period
Population: Inclusion criteria included: age ≥ 18 year old, presence of an IO placed by EMS or in the Emergency Department, and planned admission to the Medical or Surgical Intensive Care Unit. Patients were excluded if they had anticipated surgery within 12 hours of IO placement, ongoing infection at the placement site.
Measure: Number; unit: percentage of IO pressure to cuff pressu
Groups:
- Intraosseous Device Placement: Intraosseous Pressure Monitoring in Surgical Intensive Care Unit Patients
Arm/Group | Intraosseous Device Placement
Number analyzed (Participants) | 20
percentage of IO pressure to cuff pressu
  ratio as a percentage of IO SBP to cuff SBP | 34.5
  ratio as a percentage of IO DBP to cuff DBP | 40.5
  Ratio as a percentage of IO mean to cuff mean | 40.1

ADVERSE EVENTS:
Arm/Group | Intraosseous Device Placement
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes